CLINICAL TRIAL: NCT06111196
Title: A Randomized, Double-blind, Single-dose, Three-arm Parallel Group, Phase I Study to Compare the Pharmacokinetics and Safety of BAT3306 Versus KEYTRUDA® Administered in Healthy Male Subjects
Brief Title: Compare the Pharmacokinetics and Safety of BAT3306 Injection Versus KEYTRUDA® Administered in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bio-Thera Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAT-3306-001-CR
Record Dates: First submitted 2023-09-21; First posted 2023-11-01 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Healthy Male Subjects
MeSH Terms: interventions — Injections; pembrolizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- BAT3306 injection (Experimental): 100mg/4ml,intravenous injection
  Interventions: Drug: Recombinant Humanized Anti-PD-1 Monoclonal Antibody Solution for Injection
- KEYTRUDA® (EU-sourced) (Active Comparator): 100mg/4ml,intravenous injection
  Interventions: Drug: Pembrolizumab injection

INTERVENTIONS:
Drug: Recombinant Humanized Anti-PD-1 Monoclonal Antibody Solution for Injection — 100mg/4ml;single dose;intravenous injection
  Other Names: BAT3306 injection
  Arms: BAT3306 injection
Drug: Pembrolizumab injection — 100mg/4ml;single dose;intravenous injection
  Other Names: KEYTRUDA® (EU-sourced)
  Arms: KEYTRUDA® (EU-sourced)

SUMMARY:
to Compare the Pharmacokinetics and Safety of BAT3306 versus KEYTRUDA® Administered in Healthy Male Subjects

DETAILED DESCRIPTION:
A Randomized, Double-blind, Single-dose, Three-arm Parallel Group, Phase I Study to Compare the Pharmacokinetics and Safety of BAT3306 versus KEYTRUDA® Administered in Healthy Male Subjects

ELIGIBILITY:
Inclusion Criteria:

The subjects must sign the informed consent before they can start the screening procedure and entering the clinical study. They can only be included if they meet all the following criteria:

1. Adult males aged 18 to 55 years inclusive and with 18.0 to 28.0 kg/m2 body mass index (BMI) and body weight should between 50 to 85 kg（all contain boundary values）;
2. Subject is able to understand and to comply with protocol requirements, instructions, and restrictions, voluntarily agrees to participate in this study and has given a written informed consent prior to performing any of the screening procedures;
3. Physical examination, vital signs, 12-lead ECG, laboratory tests and other examination results of the subjects are normal or abnormal but with no clinical significance;
4. Non-smokers or smokers of less than 5 cigarettes per day for less than 10 years;
5. Agree to take effective contraception measures (including but not limited to: hormonal contraception, or physical contraception, or abstinence) and no sperm donation plan from the time of signing the informed consent form until 6 months after injection of study drug; 6. Must be willing and able to comply with scheduled visits, treatment plan, laboratory tests and other relevant procedures specified in this study.

Exclusion Criteria:

Subjects meeting any of the following shall not be included:

1. Have a history of and/or current clinically significant gastrointestinal (including but not limited to diverticulitis, stomach ulcers), renal, hepatic, cardiovascular, haematological， pulmonary, neurologic, metabolic (including but not limited to known diabetes mellitus), psychiatric or allergic disease excluding mild asymptomatic seasonal allergies, and other diseases that the investigator considers unsuitable for participation in this clinical study;
2. Subject with a psychiatric disorder or considered unsuitable for inclusion by the investigator (e.g., inability to understand and/or comply with study requirements or presence of any condition which, in the opinion of the investigator, would not allow safe participation in the study);
3. Previous or current clinically significant allergic disease(excluding mild asymptomatic seasonal allergy); or it is known or suspected that the subject may have allergic or hypersensitive reactions to any component of the study drug; or it is known or suspected that the subject may have allergic or hypersensitive reactions to hamster ovary cell products or other recombinant human or humanized antibodies;
4. Have a history of autoimmune disease and presence of thyroid function disorders or related history (e.g., hyperthyroidism, hypothyroidism, and other thyroid disorders);
5. Propensity for bleeding or thrombosis, or a history of non-traumatic bleeding with appropriate clinical treatment, or a history of thrombosis, or the presence of any disease that may put the subject at increased risk of bleeding or thrombosis(such as abnormal coagulation, thrombocytopenia, or INR > 1.5);
6. History of any malignancy;
7. Abnormal ECG with clinical significance (as judged by the investigator) or QT interval > 450 ms after Bazett correction (Bazett formula: Q-Tc = QT/(R-R)^0.5, where R-R denotes the interval between two R waves in s);
8. History of hypertension or systolic blood pressure > 140 mmHg or diastolic blood pressure > 90 mmHg at screening or baseline;
9. Have clinically significant chronic or acute infections at the time of screening/ enrollment; or Hepatitis B surface antigen (HBsAg) positive, or HCV, or HIV, or syphilis specific antibody test results show positive during the screening period;
10. Any prior exposure to Pembrolizumab or anti-PD-1 / L1 antibody (including monoclonal antibody, bispecific antibody and relevant target drugs);
11. Use of any biologic product within 3 months or any monoclonal antibody within 9 months prior to the study drug administration;
12. Use of prescription or over-the-counter medication within 14 days prior to study drug administration, or last dose is less than 5 half-lives from the date of administration of this study (whichever is longer);
13. Have used any herbal medicine or proprietary Chinese medicine within 14 days prior to study drug administration,;
14. Participated in another drug clinical trial within 3 months prior to study drug administration,, or intend to participate in another drug clinical trial during this study;
15. Live / attenuated or mRNA vaccine received within 4 weeks prior to study drug administration or planned to vaccination during the study;
16. Have had a major injury or previous surgical procedure or fracture within 4 weeks prior to study drug administration, or intend to have surgery during the study period;
17. Have donated blood or had a blood sample > 400ml taken as a subject within 3 months prior to screening, or plan to donate blood during the study period;
18. History of alcohol dependence or a positive screening/baseline alcohol test result;
19. Consumption of alcoholic beverages within 48h prior to study drug administration;
20. History of substance abuse, or positive drug abuse test results during the screening period;
21. Inability to comply with the study's restrictions on smoking, alcohol consumption, and concomitant medications during the study.

22. Can not stop high intensity physical exercise from the day of study drug administration till 30 days thereafter.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 59 (Actual)
Dates: Start 2023-11-05 (Actual); Primary Completion 2024-06-11 (Actual); Study Completion 2024-06-11 (Actual)

PRIMARY OUTCOMES:
CL | Day1, Day2,Day3,Day4,Day8,Day22,Day29,Day36,Day43,Day51,Day71,Day85,Day99.Day113
  Number of participants to single dose PK characteristics
Cmax | Day1, Day2,Day3,Day4,Day8,Day22,Day29,Day36,Day43,Day51,Day71,Day85,Day99.Day113
  Number of participants to Peak plasma concentration evaluation
AUC0-∞ | Day1, Day2,Day3,Day4,Day8,Day22,Day29,Day36,Day43,Day51,Day71,Day85,Day99.Day113
  Number of participants to area under the drug concentration-time curve evaluation
(AUC0-t) | Day1, Day2,Day3,Day4,Day8,Day22,Day29,Day36,Day43,Day51,Day71,Day85,Day99.Day113
  Number of participants to data point evaluation
Tmax | Day1, Day2,Day3,Day4,Day8,Day22,Day29,Day36,Day43,Day51,Day71,Day85,Day99.Day113
  Number of participants to single dose PK characteristics evaluation
t1/2 | Day1, Day2,Day3,Day4,Day8,Day22,Day29,Day36,Day43,Day51,Day71,Day85,Day99.Day113
  Number of participants to PK characteristics evaluation
Vd | Day1, Day2,Day3,Day4,Day8,Day22,Day29,Day36,Day43,Day51,Day71,Day85,Day99.Day113
  Number of participants to Single dose PK characteristics evaluation

SECONDARY OUTCOMES:
Vital signs | Day1,Day2,Day3,Day4,Day5,Day8,Day15,Day22,Day29,Day36,Day43,Day57,Day71,Day85,Day99,Day113,End of study
  Number of participants with abnormal vital signs
ECG parameters | Day1,Day2,Day5,Day15,Day43,Day113,End of study
  Number of participants with abnormal ECG readings
Laboratory tests | Day1,Day2,Day5,Day15,Day22,Day29,Day43,Day71,Day85,Day113,End of study
  Number of participants with abnormal laboratory test results
AEs, adverse events | Day1,Day2,Day3,Day4,Day5,Day8,Day15,Day22,Day29,Day36,Day43,Day57,Day71,Day85,Day99,Day113,End of study
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0
Injection site reactions | Day1,Day2, Day3,Day 4, Day5, Day15;
  Number of participants with injection site reactions
ADA antibody | Day1, Day 15, Day57, Day85, and Day113
  Number of participants to immunogenicity evaluation.
Nab positive | Day1, Day 15, Day57, Day85,Day113
  Number of participants to Immunogenicity evaluation when the ADA is positive.

CONTACTS AND LOCATIONS:
Overall Officials: Weiyong Li, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital,Tong Ji Medical College,Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No